CLINICAL TRIAL: NCT01088230
Title: The Impact of Botox® During Robotic Rehabilitation of the Wrist Following Stroke: A Double Blind, Placebo-Controlled Pilot Study
Brief Title: The Impact of Botox® During Robotic Rehabilitation of the Wrist Following Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York Presbyterian Hospital (Other)
Responsible Party: Michael O'Dell, Weill Cornell Medical College/ NewYork Presybterian Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-0904010371
Record Dates: First submitted 2010-03-11; First posted 2010-03-17 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2010-11

CONDITIONS: Stroke
Keywords: hemiparesis; robotics; stroke; Botox®; rehabilitation; wrist spasticity
MeSH Terms: conditions — Stroke; Paresis | interventions — Botulinum Toxins, Type A; Saline Solution; Fluoridation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botox® (Experimental): this group will receive an injection of botox in the wrist flexors and forearm pronators
  Interventions: Other: Botox®
- Saline (Placebo Comparator): This group will receive an injection of saline solution in the same muscle groups as the treatment group (wrist flexors and pronators).
  Interventions: Other: saline solution

INTERVENTIONS:
Other: Botox® — the treatment group will receive a one time injection of Botox® at the wrist flexors and pronators of the affected arm. Each subject will receive a standard dose of 150 units total, 50u each to the flexor carpi radialis and flexor carpi ulnaris, and 25u each for the pronator teres and pronator quadratus muscle groups.
  Other Names: botulinum toxin serotype-A
  Arms: Botox®
Other: saline solution — the control group will receive a one time injection of salt water in the flexor carpi radialis and flexor carpi ulnaris, and the pronator teres and pronator quadratus muscle groups.
  Other Names: salt water
  Arms: Saline

SUMMARY:
The purpose of this study is to see whether treating subjects for wrist rehabilitation following stroke with Botox® and robotic therapy is more effective than treatment with robotic therapy alone and no Botox®.

DETAILED DESCRIPTION:
This study will explore new ways to facilitate rehabilitation of wrist function after stroke. One of the challenges of recovery is muscle stiffness or excessive muscle tone that often limits exercise or therapy progress. Taking this into account, the investigators propose treating the wrist and forearm with a combination of a one-time Botox® injection and a 6-week robotic therapy protocol to maximize recovery.

Botox® is a drug that is injected directly into a muscle to temporarily relax the muscle. Botox® is commonly used to decrease muscle tone in tight muscles in the stroke population. Robotics therapy provides highly repetitive mass practice with visual and haptic feedback.

Subjects will be randomized to two groups. Group A will receive the Botox® injection and group B will receive a placebo saline injection. Both groups will receive the same robotics therapy protocol. Subjects and investigators will be blinded to group assignment. The investigators would like to know if there are trends between groups in a variety of outcome measures depending on what intervention they received. The investigators predict that the treatment group will have better results than the control group on the Fugl Meyer, our primary outcome measure. The investigators hope the results of this pilot study will guide development of a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* > 6 months post-stroke
* Single stroke
* Ashworth Scale of > 2 but < 4 for wrist flexors and pronators
* Able to follow multiple step directions
* Completed all active occupational therapy
* Motor strength > 1/5 at the wrist extension and supination
* Passive ROM of 0-45 degrees at wrist flexion and extension, 0-20 degrees at radial deviation, 0-20 degrees at ulnar deviation, 0-45 degrees at pronation and supination
* No Botox® injection in the wrist/forearm muscles for at least 12 months
* Naïve to robotics study protocol

Exclusion Criteria:

* Joint contracture and wrist or forearm

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change scores on Fugl Meyer- Upper Extremity Section | at baseline and discharge
  The Fugl Meyer assess quality of movement of the limb at an impairment level.

SECONDARY OUTCOMES:
Change on kinematic analysis | before injection and one week post injection
  Kinematic information is recorded during administration of the assessment mode of the InMotion 3 wrist robotic device. Movements of the wrist (flexion,extension,ulnar/radial deviation) and forearm (pronation, supination)are recorded for subsequent analysis. Kinematic parameters such as smoothness, position and velocity of movement are examined pre and post injection. The information is extracted from the robotics device and analyzed via computer programs.

CONTACTS AND LOCATIONS:
Locations (1):
- New York Presbyterian Hospital- Weill Cornell campus, New York, New York, United States

REFERENCES:
- [Background] Caty GD, Detrembleur C, Bleyenheuft C, Deltombe T, Lejeune TM. Effect of upper limb botulinum toxin injections on impairment, activity, participation, and quality of life among stroke patients. Stroke. 2009 Jul;40(7):2589-91. doi: 10.1161/STROKEAHA.108.544346. Epub 2009 Apr 30. PMID 19407231
- [Background] Fasoli SE, Fragala-Pinkham M, Hughes R, Krebs HI, Hogan N, Stein J. Robotic therapy and botulinum toxin type A: a novel intervention approach for cerebral palsy. Am J Phys Med Rehabil. 2008 Dec;87(12):1022-5. doi: 10.1097/PHM.0b013e31817fb346. PMID 18617860
- [Background] Frascarelli F, Masia L, Di Rosa G, Petrarca M, Cappa P, Castelli E. Robot-mediated and clinical scales evaluation after upper limb botulinum toxin type A injection in children with hemiplegia. J Rehabil Med. 2009 Nov;41(12):988-94. doi: 10.2340/16501977-0412. PMID 19841830
- [Background] Levy CE, Giuffrida C, Richards L, Wu S, Davis S, Nadeau SE. Botulinum toxin a, evidence-based exercise therapy, and constraint-induced movement therapy for upper-limb hemiparesis attributable to stroke: a preliminary study. Am J Phys Med Rehabil. 2007 Sep;86(9):696-706. doi: 10.1097/PHM.0b013e31813e2b4d. PMID 17709993
- See also: click here for to sign up for future stroke studies at NYPH — https://s010.med.cornell.edu/nyp/rehabmed/stroke_registry.html